CLINICAL TRIAL: NCT05909891
Title: The Effect of Education Given to Individuals with Iron Deficiency Anemia on Treatment Compliance and Fatigue
Brief Title: Treatment Adherence and Fatigue in Iron Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Hatice Polat, Assoc. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: B.30.2.ATA.0.01.00/416
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Fatigue; Adherence, Medication
Keywords: fatigue; education; anemia; adherence
MeSH Terms: conditions — Fatigue; Medication Adherence; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Patient selection will be made according to the planned randomization after examining the inclusion and exclusion criteria.
  Introductory Form, Morisky Scale and Fatigue Scale will be applied to the individuals in the experimental group included in the study. The same forms will be applied to the patients included in the control group. Individuals in the control group will be followed up by the hospital routinely.
  In addition to the routine follow-ups for the patients in the experimental group, the training material created by the researchers will be individually presented as an average of 35-40 minutes, and a session will be given in the form of mutual question and answer. After the training, a sample booklet, which is the training material, will be given to the patient as a reminder.
  Adaptation and fatigue tests will be re-applied at the first control of the patients after the training.
  Interventions: Other: Patient training
- Control Group (No Intervention)

INTERVENTIONS:
Other: Patient training — A training booklet will be created by scanning the literature on iron deficiency anemia. The training booklet will be evaluated in terms of content and readability, according to the DISCERN measurement tool, while obtaining expert opinion.
  The training period will be at least 35-40 minutes, taking into account the educational status of the patient and explaining the importance of compliance with the treatment. After the training, when the patients come to the routine check-ups in the 1st and 2nd months, the level of compliance with the treatment and the fatigue of the patients will be evaluated.
  Arms: Experimental Group

SUMMARY:
Iron Deficiency Anemia is an important health problem. Iron deficiency anemia constitutes half of the anemia seen in the world, and children and women constitute the group with iron deficiency anemia in our country. The treatment is iron replacement by oral or parenteral route. Due to the side effects of the drugs given in the treatment, the patients have difficulty in adapting to the treatment and there is a change in their fatigue levels. It is thought that the education given to the patients will increase their compliance with the treatment. It is thought that patients' hospital admissions and fatigue levels may change in the failure to comply with the treatment.

In this study, the effect of the education given on the treatment compliance and fatigue of the patients will be investigated. This research will help patients with iron deficiency anemia whether they need education, the importance of treatment compliance and their fatigue levels.

DETAILED DESCRIPTION:
Iron Deficiency Anemia (DEA) is one of the acquired anemia, which is seen as a result of insufficient intake of iron necessary for the body or rapid decrease in iron stores. It is the most common anemia in the world and constitutes 50% of anemias. It is stated that the incidence is increasing in low-income societies. In studies on adults, the frequency of IDA is around 20%, and it is most commonly seen in women due to pregnancy and menstruation.

The aim of the "Turkey Like Iron" program, which was started in our country in 2004, is to try to prevent iron deficiency anemia as new generations are the adults of the future. The most common findings in patients with iron deficiency anemia are fatigue, weakness, activity intolerance, hair loss and thinning, thinning-breaking-flattening of nails, and headache. The reason for fatigue, which is one of these symptoms, is the decrease in the amount of oxygen carried to the tissues as a result of the low hemoglobin level in the blood. Depending on the inability to carry enough oxygen to the muscles, activity intolerance occurs in people. The degree of anemia affects the severity of fatigue. The severity of fatigue also affects the person's ability to perform activities of daily living. Oral or parenteral iron replacements are used in the treatment of anemia that causes fatigue and activity intolerance. However, some side effects may be seen in patients due to the use of oral iron drugs. These side effects are stated as tooth discoloration, nausea, vomiting, indigestion, constipation, diarrhea, and darkening of stool color. Patients cannot continue treatment due to these side effects. Trainings given to patients to increase adherence to treatment can be effective in coping with the treatment process and side effects. It is stated that the symptoms experienced by the patients who continue the treatment will decrease in a short time such as 1 month. However, it was stated by the experts that the treatment should be continued for 3-6 months in order to replace the iron stores. When the increase in the hemoglobin values of the patients who continue the treatment and the oxygen carried to the tissues reach a sufficient level, the symptoms such as fatigue and activity intolerance will decrease and disappear over time.

Considering the authorities and responsibilities of the nursing profession, one of the most important is to provide training in line with the needs of the patient and their relatives. Nurses provide training to individuals in order to protect and improve the health of the individual, family and society, and to gain the right health behaviors to improve in case of illness. From past to present, training given to patients by healthcare professionals increases patients' adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Orientation to person, place and time
2. Having no problems communicating
3. To voluntarily agree to participate in the research
4. Being diagnosed with iron deficiency anemia
5. Being between the ages of 18-65
6. Being able to read and write
7. Receiving oral iron medication for at least 1 month
8. Those with low Morisky scale motivation score

Exclusion Criteria:

1. Individuals under the age of 18
2. Foreign nationals
3. Those with maling disease
4. Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Morisky Medication Adherence Scale (MMAS 4) | avarage of six mounth
  The scale was developed in 1986 by Morisky et al. to evaluate adherence to antihypertensive drug treatment. The validity and reliability study of the Morisky Adherence to Medication Scale, which is used in many studies for chronic diseases, was conducted by Yılmaz (2004) for our country to measure adherence to antipsychotic treatment. Muslu used this scale to evaluate adherence to treatment in schizophrenia patients in 2010. The scale has a 4-question design that can evaluatethe motivation and knowledge levels separately to evaluate adherence to long-term drug treatment in chronic diseases. The questions of the scale are answered as "Yes/No", and "Yes" is calculated as "0" points and "No" as "1" points. The highest total score obtained from the scale is "4", and as the score increases, treatment adherencealso increases. The score obtained from the scale indicates adherence to treatment as 0-1 = Low level, 2-3 = Moderate level, and 4 = High
Visual Similarity Scale for Fatigue | avarage of six mounth
  The Turkish validity and reliability scale was made by Yurtsever, and it was created by Lee et al. (1990) in 1990. The scale consists of 18 items, fatigue (1. 2. 3. 4. 5. 11. 12. 13. 14. 15. 16. 17. and 18. items) and energy level (6. 7. 8. 9 and 10. items) consists of sub-dimensions. There are 10 cm lines in each statement of the scale, and there is a positive statement at one end of the line and a negative statement at the other. These statements are scored between 0 and 10. The items of the fatigue subscale range from the most positive to the most negative, while the items of the energy subscale range from the most negative to the most positive. An increase in the fatigue subscale score indicates an increase in the severity of fatigue, and an increase in the energy subscale score indicates an increase in energy. Getting a high score on the fatigue questions and a low score on the energy questions indicate that the severity of fatigue is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] Houston BL, Hurrie D, Graham J, Perija B, Rimmer E, Rabbani R, Bernstein CN, Turgeon AF, Fergusson DA, Houston DS, Abou-Setta AM, Zarychanski R. Efficacy of iron supplementation on fatigue and physical capacity in non-anaemic iron-deficient adults: a systematic review of randomised controlled trials. BMJ Open. 2018 Apr 5;8(4):e019240. doi: 10.1136/bmjopen-2017-019240. PMID 29626044
- [Background] Warner MJ, Kamran MT. Iron Deficiency Anemia. 2023 Aug 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448065/ PMID 28846348
- [Background] Auerbach M, Adamson JW. How we diagnose and treat iron deficiency anemia. Am J Hematol. 2016 Jan;91(1):31-8. doi: 10.1002/ajh.24201. Epub 2015 Nov 17. PMID 26408108